CLINICAL TRIAL: NCT02738671
Title: The Cross-sectional and Longitudinal Study of Relationship Between Diabetes and Cognitive Impairment by Olfactory Function Assessment and Functional MRI in Obese and Normal Weight Diabetic Patients
Brief Title: Relationship Between Diabetes and Cognitive Impairment Based on Olfactory Function Assessment and Functional MRI
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: ZZ2016
Record Dates: First submitted 2016-02-25; First posted 2016-04-14 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2016-10

CONDITIONS: Diabetes Mellitus; Cognitive Impairment; Obesity
Keywords: functional MRI; olfactory function; bariatric surgery
MeSH Terms: conditions — Diabetes Mellitus; Cognitive Dysfunction; Obesity | interventions — Mental Status and Dementia Tests; Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Type 1 Diabetes Mellitus: These T1DM patients have late diabetes onset.(latent autoimmune diabetes in adult, LADA)
  Interventions: Behavioral: Cognitive assessment; Other: functional magnetic resonance imaging; Other: olfactory function measurement
- Type 2 Diabetes Mellitus: A subgroup of these T2DM patients are obesity patients who will have the bariatric surgery. These obese T2DM subjects will undergo a physical exam, cognitive and olfactory test as well as structural and functional brain MRI at baseline and 6 months after their surgery.
  Interventions: Behavioral: Cognitive assessment; Other: functional magnetic resonance imaging; Other: olfactory function measurement; Procedure: bariatric surgery
- Control: A subgroup of these non-diabetic people are obesity patients who will have the bariatric surgery. These obese subjects will undergo a physical exam, cognitive and olfactory test as well as structural and functional brain fMRI at baseline and 6 months after their surgery.
  Interventions: Behavioral: Cognitive assessment; Other: functional magnetic resonance imaging; Other: olfactory function measurement; Procedure: bariatric surgery

INTERVENTIONS:
Behavioral: Cognitive assessment
Other: functional magnetic resonance imaging
  Other Names: fMRI
Other: olfactory function measurement
Procedure: bariatric surgery — Only a subgroup of the subjects will have the bariatric surgery.
  Groups: Control; Type 2 Diabetes Mellitus

SUMMARY:
The purpose of this study is to explore the relationship between diabetes and cognitive impairment by olfactory function assessment and functional MRI.

DETAILED DESCRIPTION:
Previous research has shown both obesity and diabetes are associated with an increased risk of cognitive impairment. Meanwhile, olfactory impairment is associated with incident (amnestic mild cognitive impairment) aMCI and progression from aMCI to (Alzheimer disease) AD dementia. On one hand, in the cross-sectional study, biometric measurements, cognitive assessment, olfactory function and fMRI results are analysed to explore the differences among T1DM patients, T2DM patients and non-diabetic people . One the other hand, in the longitudinal study, changes in olfactory function and fMRI results in diabetic and non-diabetic obese patients both at baseline and 6 months after their bariatric surgery are collected to investigate whether better glucose and weight control benefit brain function.

ELIGIBILITY:
Inclusion Criteria:

1. Have a certain level of education (at least 6 years), able to complete the cognitive assessment;
2. Disease duration >1 year.

Exclusion Criteria:

1. Control participants would be excluded if they had a fasting blood glucose level >7.0 mmol/L; glucose level> 7.8 mmol/L after oral glucose tolerance test (OGTT);
2. Montreal Cognitive Assessment (MoCA,Beijing edition) score of < 20;
3. History of neurologic or psychological illness;
4. History of cardiovascular or cerebrovascular disease;
5. Abnormal results of thyroid hormones, vitamin B12, and folate.
6. Metal implants, unable to complete the MR examinations or evidence of cortical infarcts, hemorrhage, or structural brain disease other than atrophy, lacunes, or white matter lesions;
7. Left-handed;
8. Partial or complete olfactory dysfunction associated with sinusitis,allergic rhinitis, and deviated nasal septum.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: T1DM(latent autoimmune diabetes in adult,LADA) and T2DM patients.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Participants' personal information | 1 day
  Self-reported information(education in years)
Glycaemic control measured by blood test. | 1 day
  HbA1c
Physical assessments. | 1 Day
  BMI(body mess index) in kg/m^2
Olfactory threshold test | 1 day
  Olfactory threshold test:
  The same odor with 2 different concentrations are given to the participant each time to find out which one is more intense. (Olfactory software will analyse and give threshold score depending on participant's choice.)
Olfactory memory test: | 1 day
  PART A: Participants are shown 4 pictures for each odor(10 odors in total). They select what they sniffed.
  10 minutes break.
  PART B: Participants sniff 20 different odors , 10 of which are same odors in PART A. They select the picture and figure out whether the odor is old or new.
Montreal Cognitive Assessment (MoCA) | 1 Day
  The MoCA is a cognitive screening test designed to assist Health Professionals in detection of mild cognitive impairment.
Functional MRI of the brain tracking testing. | 1day

SECONDARY OUTCOMES:
Change form baseline Glycaemic control measured by blood test. | 6 months after the bariatric surgery (for diabetic and non-diabetic obese patients)
  HbA1c
Change from baseline Functional magnetic resonance imagine | 6 months after the bariatric surgery (for diabetic and non-diabetic obese patients)

CONTACTS AND LOCATIONS:
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhao Q, Maimaitiaili S, Bi Y, Li M, Li X, Li Q, Shen X, Wu M, Fu L, Zhu Z, Zhang X, Chen J, Hu A, Zhang Z, Zhang W, Zhang B. Brain Iron Deposition Alterations in Type 2 Diabetes Mellitus Patients With Mild Cognitive Impairment Based on Quantitative Susceptibility Mapping. J Diabetes. 2025 Jan;17(1):e70052. doi: 10.1111/1753-0407.70052. PMID 39843980
- [Derived] Miao Y, Wang J, Zhang B, Zhang W, Xu X, Hou Y, Ding Q, Yu C, Zhang Z, Bi Y, Zhu D. Altered brain spontaneous and synchronization activity in latent autoimmune diabetes in adults: A resting-state functional MRI study. Diabetes Metab Res Rev. 2023 Jan;39(1):e3587. doi: 10.1002/dmrr.3587. Epub 2022 Nov 7. PMID 36306532
- [Derived] Zhang W, Gao C, Qing Z, Zhang Z, Bi Y, Zeng W, Zhang B. Hippocampal subfields atrophy contribute more to cognitive impairment in middle-aged patients with type 2 diabetes rather than microvascular lesions. Acta Diabetol. 2021 Aug;58(8):1023-1033. doi: 10.1007/s00592-020-01670-x. Epub 2021 Mar 22. PMID 33751221
- [Derived] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Zhang W, Zhu D, Bi Y. Olfactory Dysfunction Mediates Adiposity in Cognitive Impairment of Type 2 Diabetes: Insights From Clinical and Functional Neuroimaging Studies. Diabetes Care. 2019 Jul;42(7):1274-1283. doi: 10.2337/dc18-2584. Epub 2019 May 21. PMID 31221697